CLINICAL TRIAL: NCT01345942
Title: A Randomized, Open Label, Single Dose, Two Period, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of RO5428029 Following Oral Administration in Healthy Subjects
Brief Title: A Study on the Effect of Food on the Pharmacokinetics of RO5428029 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: PP25583
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (2):
- A food (Experimental)
  Interventions: Drug: RO5428029
- B without food (Experimental)
  Interventions: Drug: RO5428029

INTERVENTIONS:
Drug: RO5428029 — Single oral dose

SUMMARY:
This open label, two period, crossover study will evaluate the safety and the effect of food on the pharmacokinetics of RO5428029 in healthy volunteers. In a crossover design, healthy subjects will be randomized to receive a single oral dose of RO5428029 with or without food, with a washout period of at least 7 days between dosing and a follow-up of 7 to 10 days after last dose. Anticipated time on study will be up to 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 to 60 years of age inclusive
* Body mass index (BMI) between 18 and 29.9 kg/m2, inclusive, and a minimum weight of 45 kg
* Female subjects must be surgically sterile or post-menopausal
* Male subjects and their partners of child-bearing potential must use 2 methods of contraception (one of which a barrier method) for the duration of the study and for at least 70 days after the last dose

Exclusion Criteria:

* Pregnant or lactating women, and male partners of women who are pregnant or lactating
* Women with reproductive potential
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard units per day on average; alcohol consumption will be prohibited at least 48 hours before screening
* Positive test for drugs of abuse
* History or symptoms of any significant disease
* Positive for HIV, hepatitis B or hepatitis C infection
* Participation in an investigational drug or device study within 3 months prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of food on pharmacokinetics (plasma concentrations) of RO5428029 following oral administration | 72 hours

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- San Antonio, Texas, United States